CLINICAL TRIAL: NCT01797770
Title: A Randomised Controlled Trial On Mechanical Bowel Preparation Versus No Mechanical Bowel Preparation In Elective Laparoscopic Surgery For Left Sided Colonic Tumours
Brief Title: Trial on Mechanical Bowel Preparation in Laparoscopic Colorectal Surgery
Acronym: MBP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: PVS Memorial Hospital (Other)
Responsible Party: Principal Investigator, Dr Prakash K, Chief GI Surgeon, PVS Memorial Hospital
Other Study IDs: PVS2
Record Dates: First submitted 2012-09-16; First posted 2013-02-22 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Rectal Cancer; Colon Cancer
Keywords: mechanical bowel preparation; Colon Cancer
MeSH Terms: conditions — Rectal Neoplasms; Colonic Neoplasms | interventions — Polyethylene Glycols; preparation No. 012074

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mechanical bowel preperation: mechanical bowel preparation with polyethylene glycol one day prior to surgery
  Interventions: Drug: polyethylene glycol; Other: No Preparation

INTERVENTIONS:
Drug: polyethylene glycol — mechanical bowel preparation with polyethylene glycol one day prior to surgery
Other: No Preparation — No laxatives or bowel preparation

SUMMARY:
This is a Randomized trial on Mechanical Bowel Preparation in Laparoscopic Colorectal Surgery. In this trial patients with left sided colon and rectal tumors were randomized to receive mechanical bowel preparation or no preparation to assess postoperative complications and outcome

DETAILED DESCRIPTION:
In this prospective randomized trial,patients were randomized to receive mechanical bowel preparation or no preparation to assess postoperative complications and outcome following elective laparoscopic surgery for left sided colon and rectal tumors. Randomization is done from the out -patient department at the time of admission, using random numbers from a computer generated list from a sealed envelope method.

Patients who did not have mechanical bowel preparation had a normal meal on the day before the operation. Those who did were given a fluid diet, and mechanical bowel preparation with polyethylene glycol one day prior to surgery.

Both groups will have the scheduled laparoscopic colonic resections. Use of diverting stoma is left to the discretion of the operating surgeon. Cases that needed a diverting stoma, will be analyzed separately.

ELIGIBILITY:
Inclusion Criteria:

* left sided colonic and rectal tumors
* eligible for elective laparoscopic surgery

Exclusion Criteria:

* Patients with intestinal obstruction or perforation.
* patients with T4b tumors.
* metastatic tumors
* patients with multiple previous abdominal surgeries

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Randomized open label study to assess effect of mechanical bowel preparation in elective laparoscopic surgery for left sided colon tumours
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
anastomotic leak | 30 days
  clinical/drain/radiological leak

SECONDARY OUTCOMES:
surgical site infection | 14 days
  superficial and deep surgical site infection
Intraoperative parameters assessment | 1 day
  intraoperative assessment of tumor site, extend, operative time, intraoperative contamination
bowel recovery | 30 days
  Day of passage of flatus or faeces
drain removal | 30 days
  postoperative day of drain removal
Re-exploration | 30 days
  Any intervention radiological or surgical due to procedure related complications
Hospital stay | 30 days
  postoperative hospital stay
Readmission | 30days
  admission to hospital after discharge due to any reasons

CONTACTS AND LOCATIONS:
Locations (1):
- PVS Memorial Hospital, Kochi, Kerala, India

REFERENCES:
- [Background] Contant CM, Hop WC, van't Sant HP, Oostvogel HJ, Smeets HJ, Stassen LP, Neijenhuis PA, Idenburg FJ, Dijkhuis CM, Heres P, van Tets WF, Gerritsen JJ, Weidema WF. Mechanical bowel preparation for elective colorectal surgery: a multicentre randomised trial. Lancet. 2007 Dec 22;370(9605):2112-7. doi: 10.1016/S0140-6736(07)61905-9. PMID 18156032
- [Background] Bucher P, Gervaz P, Soravia C, Mermillod B, Erne M, Morel P. Randomized clinical trial of mechanical bowel preparation versus no preparation before elective left-sided colorectal surgery. Br J Surg. 2005 Apr;92(4):409-14. doi: 10.1002/bjs.4900. PMID 15786427
- [Background] Guenaga KF, Matos D, Wille-Jorgensen P. Mechanical bowel preparation for elective colorectal surgery. Cochrane Database Syst Rev. 2011 Sep 7;2011(9):CD001544. doi: 10.1002/14651858.CD001544.pub4. PMID 21901677
- [Background] van't Sant HP, Weidema WF, Hop WC, Lange JF, Contant CM. Evaluation of morbidity and mortality after anastomotic leakage following elective colorectal surgery in patients treated with or without mechanical bowel preparation. Am J Surg. 2011 Sep;202(3):321-4. doi: 10.1016/j.amjsurg.2010.10.018. PMID 21871987